CLINICAL TRIAL: NCT05671302
Title: Walk Together: A Family-Based Intervention for Hypertension In African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sarah Woods, ASSOC PROFESSOR - Family Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0568; R21MD017658-01 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2023-01-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Family Relations
Keywords: Family support; Integrated health care systems; Healthy lifestyle; Community-based participatory research; African Americans
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Walk Together (Experimental): Walk Together involves four sessions delivered in patients' primary care clinic over approximately two months. Sessions are dyadic (i.e., all sessions include the patient and a family support person), last 30-90 minutes, and are delivered by a trained family therapist. The intervention is a culturally-response, family-based intervention that is strengths-based and includes components of integrative behavioral couples therapy and motivational interviewing. The goals of the intervention are to (a) optimize family support and communication, (b) improve hypertension knowledge, (c) enhance self-management goal-setting, and (d) increase shared problem-solving to address self-management adherence barriers. Environmental barriers to adherence are also addressed consistent with standard care.
  Interventions: Behavioral: Walk Together

INTERVENTIONS:
Behavioral: Walk Together — Receive training in the use of a study-provided blood pressure cuff and hypertension education; engage in hypertension self-management goal-setting; identify barriers to self-management adherence and utilize shared problem-solving to address barriers; connect to existing clinic resources to address environmental barriers; promote relationship strengths; practice communication and behavioral skills to address relationship concerns; engage family in support of patient self-management goals.

SUMMARY:
The goal of this study is to determine the feasibility and acceptability of a novel family-based hypertension self-management intervention, Walk Together, adapted from an existing empirically-supported dyadic intervention, for implementation in primary care.

DETAILED DESCRIPTION:
Hypertension is the driving risk factor for disparities in mortality and life expectancy between African Americans and Whites. Hypertension self-management (including blood pressure monitoring, diet, exercise, and other lifestyle changes) is critical for improving hypertension control, and prior interventions have emphasized promoting patient-level behavior change to improve self-management adherence. Though family members make substantial contributions to hypertension self-management for African Americans, family support is consistently underutilized by current hypertension self-management interventions. Family-based interventions for improving self-management are effective for other chronic conditions, including for African Americans. Evidence has demonstrated the unique and important role of family support in African Americans' hypertension management, and African Americans' preferences for the direct involvement of family in hypertension interventions. The study team will develop a family-based hypertension self-management intervention ("Walk Together") for African Americans with uncontrolled hypertension that integrates community-based participatory perspectives in the specifics of the intervention. The study team will pilot trial the culturally-adapted intervention in a primary care setting in order to examine the feasibility and acceptability of the Walk Together protocol.

ELIGIBILITY:
Inclusion Criteria:

* Black or African American
* Age 18 to 75
* Two blood pressure values ≥ 130/ ≥ 80 in 12 months prior
* Available family support person to join the intervention who agrees to participate
* English-speaking

Exclusion Criteria:

* Family support person is under the age of 18
* Documented cognitive impairment in patient's medical record
* Presence of severe psychiatric condition (i.e., current psychotic disorder or suicidality)
* Participation in prior hypertension health education intervention
* Prior participation in formative study activities (i.e., study focus groups)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention as measured by the number of participants accrued | 11 months
  Feasibility of intervention is measured by the number of participants accrued or consented and ready to participate to meet the recruitment goal of 30 dyads
Feasibility of intervention as measured by the rate of refusal among eligible patients/family members | 11 months
  Feasibility of intervention is measured by the rate of refusal among eligible patients/family members which is the number of participants refusing to consent
Adherence to the intervention as measured by the proportion of dyads successfully completing the four intervention components | 11 months
  Adherence to the intervention as measured by the proportion of dyads successfully completing the four intervention components
Adherence to the intervention as measured by the proportion of participants completing post-treatment assessments | 11 months
  Adherence to the intervention as measured by the proportion of participants completing post-treatment assessment
Attrition as measured by the proportion of consented participants who dropped out of the entire study | 11 months
  Attrition is defined as measured by the proportion of consented participants who dropped out of the entire study. If the dropout rate is more than 20% then it will be considered as attrition
Acceptability of intervention as measured by 8-item Client Satisfaction Questionnaire | Protocol completion (approx. 24 months)
  Acceptability of intervention is measured by 8-item Client Satisfaction Questionnaire. Possible scores range from 8 to 32, with higher values indicating higher satisfaction

SECONDARY OUTCOMES:
Family relationship quality as measured by the FACES-IV Short Form at Baseline | Baseline
  Family relationship quality is measured by the Family Adaptability and Cohesion Scale IV (FACES-IV) Short Form. Possible scores range from 1-5 where higher scores indicate better outcome.
Family relationship quality as measured by the FACES-IV Short Form at following session 3 | Following session 3 (Feedback Session, approx. 2-3 weeks after Baseline)
  Family relationship quality is measured by the Family Adaptability and Cohesion Scale IV (FACES-IV) Short Form. Possible scores range from 1-5 where higher scores indicate better outcome.
Family relationship quality as measured by the FACES-IV Short Form at following session 4 | Following session 4 (Booster Check-in session, approx. 7-8 weeks after Baseline)
  Family relationship quality is measured by the Family Adaptability and Cohesion Scale IV (FACES-IV) Short Form. Possible scores range from 1-5 where higher scores indicate better outcome.
Family relationship quality as measured by the Chronic Illness Resources Survey at Baseline | Baseline
  Family relationship quality is measured by the Chronic Illness Resources Survey. Possible scores range from 1-5 where higher scores indicate better outcome.
Family relationship quality as measured by the Chronic Illness Resources Survey following session 3 | Following session 3 (Feedback Session, approx. 2-3 weeks after Baseline)
  Family relationship quality is measured by the Chronic Illness Resources Survey. Possible scores range from 1-5 where higher scores indicate better outcome.
Family relationship quality as measured by the Chronic Illness Resources Survey following session 4 | Following session 4 (Booster Check-in session, approx. 7-8 weeks after Baseline)
  Family relationship quality is measured by the Chronic Illness Resources Survey. Possible scores range from 1-5 where higher scores indicate better outcome.
Health knowledge as measured by the Hypertension (HTN) Evaluation of Lifestyle and Management Knowledge scale at Baseline | Baseline
  Health knowledge is measured by the HTN Evaluation of Lifestyle and Management Knowledge scale. Possible scores range from 0-14 where higher scores indicate better health knowledge.
Health knowledge as measured by the Hypertension (HTN) Evaluation of Lifestyle and Management Knowledge scale following session 3 | Following session 3 (Feedback Session, approx. 2-3 weeks after Baseline)
  Health knowledge is measured by the HTN Evaluation of Lifestyle and Management Knowledge scale. Possible scores range from 0-14 where higher scores indicate better health knowledge.
Health knowledge as measured by the Hypertension (HTN) Evaluation of Lifestyle and Management Knowledge scale following session 4 | Following session 4 (Booster Check-in session, approx. 7-8 weeks after Baseline)
  Health knowledge is measured by the HTN Evaluation of Lifestyle and Management Knowledge scale. Possible scores range from 0-14 where higher scores indicate better health knowledge.
HTN self-management as measured by the HTN Self-Care Activity Level Effects measure at Baseline | Baseline
  HTN self-management is measured by the HTN Self-Care Activity Level Effects measure. The Hypertension Self-Care Activity Level Effects (H-SCALE) questionnaire assesses adherence to hypertension medication (possible subscale scores range from 0-21), physical activity engagement (possible subscale scores range from 0-14), eating a healthy diet (possible subscale scores range from 0-77), alcohol intake (possible subscale scores range from 0-1), tobacco exposure (possible subscale scores range from 0-14), and weight management (possible subscale scores range from 10-50). Possible cumulative adherence (index) scores range from 0-6 where higher scores indicate better adherence.
HTN self-management as measured by the HTN Self-Care Activity Level Effects measure at Baseline | Following session 3 (Feedback Session, approx. 2-3 weeks after Baseline)
  HTN self-management is measured by the HTN Self-Care Activity Level Effects measure. The Hypertension Self-Care Activity Level Effects (H-SCALE) questionnaire assesses adherence to hypertension medication (possible subscale scores range from 0-21), physical activity engagement (possible subscale scores range from 0-14), eating a healthy diet (possible subscale scores range from 0-77), alcohol intake (possible subscale scores range from 0-1), tobacco exposure (possible subscale scores range from 0-14), and weight management (possible subscale scores range from 10-50). Possible cumulative adherence (index) scores range from 0-6 where higher scores indicate better adherence.
HTN self-management as measured by the HTN Self-Care Activity Level Effects measure at Baseline | Following session 4 (Booster Check-in session, approx. 7-8 weeks after Baseline)
  HTN self-management is measured by the HTN Self-Care Activity Level Effects measure. The Hypertension Self-Care Activity Level Effects (H-SCALE) questionnaire assesses adherence to hypertension medication (possible subscale scores range from 0-21), physical activity engagement (possible subscale scores range from 0-14), eating a healthy diet (possible subscale scores range from 0-77), alcohol intake (possible subscale scores range from 0-1), tobacco exposure (possible subscale scores range from 0-14), and weight management (possible subscale scores range from 10-50). Possible cumulative adherence (index) scores range from 0-6 where higher scores indicate better adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Woods, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Family Medicine Clinic at Texas Health Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woods SB, Hiefner AR, Udezi V, Slaughter G, Moore R, Arnold EM. 'They should walk with you': the perspectives of African Americans living with hypertension and their family members on disease self-management. Ethn Health. 2023 Apr;28(3):373-398. doi: 10.1080/13557858.2022.2040958. Epub 2022 Feb 28. PMID 35227154